CLINICAL TRIAL: NCT00941603
Title: A Phase 2 Randomized, Double-Blind, Dose-Response Efficacy and Safety Study of SCH 900271 Compared to Placebo in Subjects With Primary Hypercholesterolemia (Familial and Nonfamilial) or Mixed Hyperlipidemia
Brief Title: Phase 2 Dose-Ranging Efficacy and Safety Trial of SCH 900271 in Participants With Primary Hypercholesterolemia or Mixed Hyperlipidemia (P05675)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05675; MK-8271-004 (Other: Merck protocol number)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Primary Hypercholesterolemia; Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SCH 900271 15 mg (Experimental): Participants receive SCH 900271 15 mg tablet and placebo tablet once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: SCH 900271 15mg
- SCH 900271 10 mg (Experimental): Participants receive SCH 900271 10 mg tablet and placebo tablet once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: SCH 900271
- SCH 900271 5 mg (Experimental): Participants receive SCH 900271 5 mg tablet and placebo tablet once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: SCH 900271
- SCH 900271 2.5 mg (Experimental): Participants receive SCH 900271 2.5 mg tablet and placebo tablet once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: SCH 900271
- SCH 900271 1 mg (Experimental): Participants receive SCH 900271 1 mg tablet and placebo tablet once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: SCH 900271
- Placebo (Placebo Comparator): Participants receive two placebo tablets once daily in the morning with water in a fasted state for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 900271 15mg — oral tablets; SCH 900271 - 15 mg taken once daily for 8 weeks
  Arms: SCH 900271 15 mg
Drug: SCH 900271 — oral tablets; SCH 900271 10 mg taken once daily for 8 weeks
  Arms: SCH 900271 10 mg
Drug: SCH 900271 — oral tablets; SCH 900271- 5 mg taken once daily for 8 weeks
  Arms: SCH 900271 5 mg
Drug: SCH 900271 — oral tablets; SCH 900271- 2.5 mg taken once daily for 8 weeks
  Arms: SCH 900271 2.5 mg
Drug: SCH 900271 — oral tablets; SCH 900271- 1 mg taken once daily for 8 weeks
  Arms: SCH 900271 1 mg
Drug: Placebo — oral tablets; placebo administered once daily during the 5-week single-blind placebo run-in and diet stabilization period and during the 8 week double-blind treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of SCH 900271 compared to placebo on the reduction of low-density lipoprotein cholesterol (LDL-C) from baseline to 8 weeks of treatment in participants with primary hypercholesterolemia (familial and nonfamilial) or mixed hyperlipidemia. The study will also evaluate the effect of SCH 900271 on non-high density lipoprotein cholesterol (non-HDL-C) and various other lipids and lipoproteins. The safety of SCH 900271 in this participant population will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults of either sex 18 to 75 years of age, inclusive, with a diagnosis of primary hypercholesterolemia (familial and nonfamilial) or mixed hyperlipidemia (increased LDL-C and triglycerides [TG])
* must be free of any clinically significant disease, other than primary hypercholesterolemia or mixed hyperlipidemia that would knowingly interfere with study evaluations
* must be willing to adhere to dietary recommendations, protocol requirements, and provide written informed consent

Exclusion Criteria:

The participant will be excluded from entry if ANY of the criteria listed below are met:

* use of any investigational drug within 30 days of study entry
* female of childbearing potential or lactating
* postmenopausal (or perimenopausal) woman who is currently experiencing hot flashes (e.g. within 30 days of study entry
* homozygous familial hypercholesterolemia
* congestive heart failure New York Heart Association (NYHA) Class III or IV
* uncontrolled hypertension on or off therapy
* cardiac arrhythmia requiring medication
* clinical atherosclerotic disease that confers high risk for coronary heart disease (CHD) events (e.g. clinical CHD, symptomatic carotid artery disease, peripheral arterial disease, abdominal aortic aneurysm)
* Type 1 Diabetes Mellitus
* Type 2 Diabetes Mellitus
* history of mental instability, drug/alcohol abuse or who has been treated or is being treated for severe psychiatric illness, which in the opinion of the investigator, may interfere with optimal participation in the study
* gastrointestinal ulcer within 3 months of study entry
* history of coagulopathy
* history of gout
* known active or chronic hepatic or biliary disease.
* known significant impairment of renal function, dysproteinemia, nephrotic syndrome, or other renal disease
* body mass index >40 kg/m^2
* taking non-steroidal anti-inflammatory drugs (NSAIDS) (acetaminophen and cyclooxygenase-2 [COX-2] inhibitors are allowed)
* taking more than 100 mg aspirin per day
* being treated with corticosteroids (oral, intramuscular, or intravascular)
* more than 3 alcoholic beverages per day or its equivalent (one drink equals 1.5 ounces of 80 proof liquor or equivalent) during study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2010-02-22 (Actual); Study Completion 2010-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05675&kw=P05675&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCH 900271 15 mg | SCH 900271 10 mg | SCH 900271 5 mg | SCH 900271 2.5 mg | SCH 900271 1 mg | Placebo
Started | 104 | 105 | 104 | 104 | 105 | 97
Completed | 93 | 89 | 99 | 100 | 101 | 94
Not Completed | 11 | 16 | 5 | 4 | 4 | 3
Not completed — Adverse Event | 10 | 15 | 5 | 1 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Did not meet protocol eligibility | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 900271 15 mg | SCH 900271 10 mg | SCH 900271 5 mg | SCH 900271 2.5 mg | SCH 900271 1 mg | Placebo | Total
Number analyzed (Participants) | 104 | 105 | 104 | 104 | 105 | 97 | 619
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (9.5) | 56.0 (10.8) | 56.1 (10.3) | 56.5 (8.7) | 57.5 (9.4) | 55.2 (9.5) | 56.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 49 | 50 | 52 | 47 | 300
  Male | 53 | 54 | 55 | 54 | 53 | 50 | 319

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Direct LDL-C at Week 8
Description: The percentage change from baseline in the participants' LDL-C was to be evaluated at study Week 8. Standard error presented below is least squares standard error.
Time Frame: Baseline and Week 8
Population: Intent-to-treat population defined as all participants who receive randomized treatment assignment, and have a baseline and at least one post-baseline LDL-C determination.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | SCH 900271 15 mg | SCH 900271 10 mg | SCH 900271 5 mg | SCH 900271 2.5 mg | SCH 900271 1 mg | Placebo
Number analyzed (Participants) | 102 | 105 | 103 | 101 | 105 | 96
Percent change | -2.0 (1.3) | -1.5 (1.3) | -4.2 (1.3) | 0.2 (1.3) | 1.2 (1.3) | 1.5 (1.4)
Statistical Analysis 1: Comparison: SCH 900271 15 mg vs Placebo; Test type: Superiority or Other; p = 0.06, ANOVA; Least-square (LS) means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -3.5, 95% CI 2-sided [-7.2 to 0.2]
Statistical Analysis 2: Comparison: SCH 900271 10 mg vs Placebo; Test type: Superiority or Other; p = 0.10, ANOVA — LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -3.1, 95% CI 2-sided [-6.7 to 0.6]
Statistical Analysis 3: Comparison: SCH 900271 5 mg vs Placebo; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Test type: Superiority or Other; p < 0.01, ANOVA; Difference in percent = -5.7, 95% CI 2-sided [-9.4 to -2.0]
Statistical Analysis 4: Comparison: SCH 900271 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.48, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -1.3, 95% CI 2-sided [-5.0 to 2.4]
Statistical Analysis 5: Comparison: SCH 900271 1 mg vs Placebo; Test type: Superiority or Other; p = 0.85, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -0.4, 95% CI 2-sided [-4.0 to 3.3]

2. Secondary Outcome: Change From Baseline in Direct Non-HDL-C at Week 8
Description: The percentage change from baseline in the participants' non-HDL-C was to be evaluated at study Week 8. Standard error presented below is least squares standard error.
Time Frame: Baseline and Week 8
Population: Intent-to-treat population defined as all participants who receive randomized treatment assignment and have a baseline and at least one post-baseline non-HDL-C determination.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | SCH 900271 15 mg | SCH 900271 10 mg | SCH 900271 5 mg | SCH 900271 2.5 mg | SCH 900271 1 mg | Placebo
Number analyzed (Participants) | 102 | 105 | 104 | 102 | 105 | 97
Percent change | -2.1 (1.2) | -2.7 (1.2) | -3.5 (1.2) | -0.5 (1.3) | 1.6 (1.2) | 0.9 (1.3)
Statistical Analysis 1: Comparison: SCH 900271 15 mg vs Placebo; Test type: Superiority or Other; p = 0.09, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -3.0, 95% CI 2-sided [-6.5 to 0.4]
Statistical Analysis 2: Comparison: SCH 900271 10 mg vs Placebo; Test type: Superiority or Other; p = 0.04, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -3.6, 95% CI 2-sided [-7.1 to -0.2]
Statistical Analysis 3: Comparison: SCH 900271 5 mg vs Placebo; Test type: Superiority or Other; p = 0.01, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -4.4, 95% CI 2-sided [-7.9 to -1.0]
Statistical Analysis 4: Comparison: SCH 900271 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.41, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = -1.4, 95% CI 2-sided [-4.9 to 2.0]
Statistical Analysis 5: Comparison: SCH 900271 1 mg vs Placebo; Test type: Superiority or Other; p = 0.68, ANOVA; LS means and LS standard errors based on ANOVA model extracting effects due to treatment, gender, and primary diagnosis; Difference in percent = 0.7, 95% CI 2-sided [-2.7 to 4.2]

ADVERSE EVENTS:
Time Frame: up to approximately 96 days (including 30 days following last dose for serious adverse events)
Description: Non-serious adverse events: treatment-emergent adverse events are reported. One participant in the SCH 900271 15 mg group was randomized but did not receive study drug. This participant was not included in the analyses of serious and non-serious adverse events.
Arm/Group | SCH 900271 15 mg | SCH 900271 10 mg | SCH 900271 5 mg | SCH 900271 2.5 mg | SCH 900271 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/103 | 1/105 | 3/104 | 0/104 | 0/105 | 0/97
Other Adverse Events (participants affected / at risk) | 41/103 | 41/105 | 19/104 | 8/104 | 14/105 | 5/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 900271 15 mg (N=103) | SCH 900271 10 mg (N=105) | SCH 900271 5 mg (N=104) | SCH 900271 2.5 mg (N=104) | SCH 900271 1 mg (N=105) | Placebo (N=97)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 900271 15 mg (N=103) | SCH 900271 10 mg (N=105) | SCH 900271 5 mg (N=104) | SCH 900271 2.5 mg (N=104) | SCH 900271 1 mg (N=105) | Placebo (N=97)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 6 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 18 (20) | 21 (24) | 8 (9) | 2 (2) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (18) | 18 (21) | 7 (7) | 2 (2) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (6) | 6 (7) | 3 (3) | 3 (3) | 2 (2)
Flushing (Vascular disorders) | 18 (19) | 14 (14) | 3 (3) | 1 (1) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.